CLINICAL TRIAL: NCT06784583
Title: A Study on Transcutaneous Vagus Nerve Stimulation in Perioperative Period of Percutaneous Coronary Intervention: A Randomized Clinical Trial
Brief Title: A Study on Transcutaneous Vagus Nerve Stimulation in Perioperative Period of Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guozhe Sun (Other)
Responsible Party: Sponsor-Investigator, Guozhe Sun, sub-investigator of Department of Cardiology in First Hospital of China Medical University, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2023]342
Record Dates: First submitted 2025-01-10; First posted 2025-01-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Hypertension
Keywords: percutaneous coronary intervention; Vagus Nerve Stimulation; perioperative blood pressure
MeSH Terms: conditions — Coronary Artery Disease; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous auricular vagus nerve stimulation (Experimental)
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- sham transcutaneous auricular vagus nerve stimulation (Sham Comparator)
  Interventions: Device: sham transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — 1. Prior to execution: Remove jewelry (such as earrings) that may interfere with the electrode placement; attach the electrodes to the tragus of the left ear; feed the wires over the right shoulder from the back of the neck, and then turn on the device.
  2. Initiate stimulation: Establish the following parameters: 200 μs pulse width, 30 Hz frequency, 0-36 mA current intensity (modify to the most appropriate stimulation intensity based on the patient's pain perception), and one-hour timing. Next, begin the stimulation.
  3. Stimulation end: After an hour, the device will be automatically switched off. And the procedure is finished.
  Arms: transcutaneous auricular vagus nerve stimulation
Device: sham transcutaneous auricular vagus nerve stimulation — 1. Prior to execution: Remove jewelry (such as earrings) that may interfere with the electrode placement; attach the electrodes to the tragus of the left ear; feed the wires over the right shoulder from the back of the neck, and then turn on the device.
  2. Initiate stimulation: Establish the following parameters: 200 μs pulse width, 30 Hz frequency, 0-36 mA current intensity (modify to the most appropriate stimulation intensity based on the patient's pain perception). Next, turn off the stimulation，and one-hour timing.
  3. Stimulation end: After an hour, the device will be removed and the procedure is finished.
  Arms: sham transcutaneous auricular vagus nerve stimulation

SUMMARY:
The goal of this clinical trial is to study the effect of transcutaneous auricular vagus nerve stimulation on perioperative blood pressure.

The main question it aims to answer is:

•Wether the transcutaneous auricular vagus nerve stimulation have advantages in perioperative blood pressure elevation.

Participants will sign an informed consent form, collaborate with data collection, and are randomly divided into two groups(1:1) to accept the intervention measures from corresponding groups. Researchers will record the perioperative blood pressure and compare intervention group with sham group to see if there is any difference in perioperative blood pressure.

DETAILED DESCRIPTION:
Sharp variations in blood pressure are more common in patients with hypertension. In non-cardiac procedures, up to 25% of patients will experience perioperative hypertension, which raises the risk of bleeding, cerebrovascular accidents, and cardiovascular events. Significant contributing factors include excessive sympathetic nerve activation, intraoperative and postoperative discomfort, and patient anxiety prior to surgery. The primary cause of perioperative hypertension is the malfunction of arterial dilatation and contraction brought on by renin-angiotensin system activation, which offers fresh approaches to perioperative blood pressure management.

Numerous research conducted in recent years have demonstrated that auricular stimulation of the vagus nerve can also have a number of effects on different parts of the brain, resulting in the regulation of the autonomic nerve balance in the heart. In healthy people, transcutaneous vagus nerve stimulation can lower cardiovascular sympathetic nerve excitability and control the sensitivity of baroreceptor reflexes, both of which are crucial for blood pressure regulation.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 70 years old, regardless of gender
* Patients with indications for coronary artery stent implantation
* hypertension history
* Voluntarily participate and sign an informed consent form

Exclusion Criteria:

* Patients with acute myocardial infarction
* Patients with heart failure of NYHA class III - IV
* Patients with atrial fibrillation (indicated by definite medical history or electrocardiogram on admission)
* Patients with a medical history of hyperthyroidism
* Patients with subclavian artery occlusion (indicated by definite medical history or a difference in systolic blood pressure of more than 20 mmHg between the two upper limbs)
* With an estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73m² on admission
* Patients with infections and fever
* Patients who are unable to cooperate due to mental and psychological disorders (such as mania, depression)
* Patients with tinnitus and vertigo
* Pregnant women or patients who are attempting to get pregnant
* Patients participating in clinical trials of other drugs or medical devices
* Patients deemed unsuitable by the researchers to participate in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure in the catheterization laboratory. | Before PCI in the catheterization laboratory
  comparation of systolic blood pressures, diastolic blood pressure and pulse between two groups in the catheterization laboratory.

SECONDARY OUTCOMES:
Incidence of perioperative hypertensive crisis | 24 hours before operation.
  Mean preoperative systolic blood pressure in the catheterization laboratory of ≥180 mmHg and/or diastolic blood pressure of ≥110 mmHg and/or temporary pharmacologic intervention for significantly elevated blood pressure 24 hours before operation.
Preoperative blood pressure difference | preoperative and the previous day's 6 o'clock
  The difference between the preoperative and the previous day's 6 o'clock blood pressure in the catheterization laboratory
Preoperative blood pressure control rate in the catheterization laboratory. | Operation day (before procedure)
  Mean preoperative blood pressure <140/90 mmHg in the catheterization laboratory was recorded as achieved;
Difference in anxiety status | Operation day ( before procedure)
  The anxiety status of subjects in the catheterization laboratory was evaluated using the Visual Analog Scale (VAS). This scale ranges from 0 to 10 points (with the minimum score of 0 and the maximum score of 10), and higher scores indicate a higher level of anxiety.
Safety evaluation | Perioperative period
  Procedure-related adverse events and device-related adverse events; the former included Major Adverse Cardiac Events (MACE) (all-cause mortality, myocardial infarction, target vessel revascularization, and stroke) and intraoperative antihypertensive medication interventions; device-related adverse events included irritation site itching and tingling, and vagal reflex.

CONTACTS AND LOCATIONS:
Overall Officials: Yingxian Sun, Principal Investigator — First Hospital of China Medical University
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China